CLINICAL TRIAL: NCT03847883
Title: Low-dose Versus Standard-dose Ateplase in Acute Ischemic Stroke ; A 4 Months Prospective Randomized Control Pilot Follow by Single Arm Standard Dose Ateplase Study.
Brief Title: Low-dose Versus Standard Dose Alteplase in Acute Ischemic Stroke , 4 Monthes Prospective Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Lumpang Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Subsai Kongsaengdao, Associated Professor, Department of Medical Services Ministry of Public Health of Thailand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rajavithi Lumphang 001 study
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Acute Stroke
Keywords: Ateplase; Intravenous recombinant tissue plasminogen activator; Acute is hemic stroke; Low-dose Ateplase; rtPa; Modified Rankin 's Scale
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Cohort A double blind Randomized controlled trial 0.6 or 0.7 or 0.9 mg/Kg Ateplase in78 patients (preliminary) Cohort B single arm standard dose 0.9 mg/kg Ateplase in 330 patients
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.6 mg/kg Ateplase (Active Comparator): Low dose 0.6 mg/kg Ateplase injection with in 4.5 Hr after onset of stroke (n = 26 in cohort A)
  Interventions: Drug: Intravenous Solution Ateplase
- 0.75 mg/kg Ateplase (Active Comparator): Low dose 0.75 mg/kg Ateplase injection with in 4.5 Hr after onset of stroke(n = 26 in cohort A)
  Interventions: Drug: Intravenous Solution Ateplase
- 0.9 mg/kg Ateplase (Active Comparator): Low dose 0.9 mg/kg Ateplase injection with in 4.5 Hr after onset of stroke(n = 26 in cohort A and n= 330 in Cohort B)
  Interventions: Drug: Intravenous Solution Ateplase

INTERVENTIONS:
Drug: Intravenous Solution Ateplase — Infusion Low dose 0.6 or 0.75 or 0.9 mg/kg Ateplase injection iv bolus 10% of total dose and infusion 90% of total dose in1 hour , with in 4.5Hr after onset of stroke

SUMMARY:
Cohort A Randomized Control trial of Ateplase 0.6, 0.75 and 0.9 mg/kg in 78 patients Cohort B single arm 0.9 mg/kg Ateplase in 330 patients Combined Cohort A and B evaluate different of death, intra-cerebral hemorrhage, numberof patient with mRS 0-1 at discharge and 3 months follow up, and other important stroke outcomes

DETAILED DESCRIPTION:
We conducted the prospective study to compare the low-dose and standard-dose rtPa and identify the important factors predicted stroke outcomes in acute stroke patient received intravenous rtPa. In Cohort A, During 2011-2012, 78 patients were randomly assigned to received intravenous rtPa 0.6 mg/kg , 0.75 mg/Kg, or 0.9 mg/Kg (1:1:1). After interim analysis during 2012-2017, in Cohort B, 330 patients were assigned to receive standard-dose rtPa 0.9 mg/kg. The good outcomes were defined as improvement of modified Rankin scale (mRS) by final score 0-1 or improvement > 4 points at discharge or 3 months follow up, absent of intracranial hemorrhage within 36 hours treatment, 90-day post-stroke survival , and short hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Acute ischemic stroke
2. Age 18 to 80 years
3. Onset of stroke symptoms with in 4.5 hours before initiation of study-drug administration
4. Stroke symptoms present for at least 30 minutes with no significant improvement before treatment

Exclusion Criteria:

1. patients with Intracranial hemorrhage
2. the symptoms of Time onset was unknown
3. Symptoms rapidly improving or only minor before start of infusion
4. Seizure at the onset of stroke
5. Stroke or serious head trauma within the previous 3 months
6. Administration of heparin within the 48 hours preceding the onset of stroke, with an activate
7. partial-thromboplastin time at presentation exceeding the upper limit of the normal range
8. Platelet count of less than 100,000 per cubic millimeter
9. Systole pressure greater than 185 mm Hg or diastole pressure greater than 110 mm Hg, or aggressive treatment intravenous medication) necessary to reduce blood pressure to these limits
10. Blood glucose less than 50 mg per deciliter or greater than 400 mg per deciliter
11. Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal
12. Oral anticoagulant treatment
13. Major surgery or severe trauma within the previous 3 months
14. Other major disorders associated with an increased risk of bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Death in 36 hours | 0-36 hours
  Number of patient die in 36 hours
Death in 3 months | 0-3 months
  Number of patient die in 3 months
Death in 4 months | 0-4 months
  Number of patient die in 4 months
Total number of patients with mRS 0-1 at discharged | 1day to <3 months
  Number of patients with mRS 0-1 at discharge 1day to 3 months interval
Total number of patients with mRS 0-1 at 3 months | At 3 months
  Number of patients with mRS 0-1 at 3 months
Number of patients with All intra-cerebral hemorrhage (ICH) at 36 hours | 0- 36 hours
  Total Intracerebral hemorrhage (ICH) including both Symptomatic ICH , and Asymptomatic ICH
Number of patients with All intra-cerebral hemorrhage (ICH) at 3 months | 0-3 months
  Total Intracerebral hemorrhage (ICH) including both Symptomatic ICH , and Asymptomatic ICH
Number of patients with All Intra-cerebral hemorrhage (ICH) at 4months | 0-4 months
  Total Intracerebral hemorrhage (ICH) including both Symptomatic ICH , and Asymptomatic ICH
Number of patients with Symptomatic Intra-cerebral hemorrhage (ICH) at 36 hours | 0-36 hours
  Total Number of patients with Symptomatic ICH need emergency surgery craniotomy or Venticulostomy drainaged or other management to reduce intracranial pressure such as intubation with mechanical ventilator or hyperosmolar drug administration
Number of patients with Symptomatic Intra-cerebral hemorrhage (ICH) at 4 months | 0-4 months
  Total Number of patients with Symptomatic ICH need emergency surgery craniotomy or Venticulostomy drainaged or other management to reduce intracranial pressure such as intubation with mechanical ventilator or hyperosmolar drug administration
Number of patients with Asymptomatic Intra-cerebral hemorrhage (ICH) 36 hours | 0-36 hours
  Total Number of patients with Asymptomatic ICH wich no need emergency surgery craniotomy or Venticulostomy drainaged or other management to reduce intracranial pressure such as intubation with mechanical ventilator or hyperosmolar drug administration
Number of patients with Asymptomatic Intra-cerebral hemorrhage (ICH) 3 months | 0-3 months
  Total Number of patients with Asymptomatic ICH wich no need emergency surgery craniotomy or Venticulostomy drainaged or other management to reduce intracranial pressure such as intubation with mechanical ventilator or hyperosmolar drug administration
Number of patients with Asymptomatic Intra-cerebral hemorrhage (ICH) 4 months | 0-4 months
  Total Number of patients with Asymptomatic ICH wich no need emergency surgery craniotomy or Venticulostomy drainaged or other management to reduce intracranial pressure such as intubation with mechanical ventilator or hyperosmolar drug administration

SECONDARY OUTCOMES:
Good stroke outcomes | 0-4 months
  Total number of patients with "good outcomes" were defined as number of patients with this any one item criteria
  1. improvement of modified Rankin scale (mRS) by final score 0-1
  2. mRS improvement > 4 points at discharge or 3 months follow up, And must full fill all of this criteria
  1) absent of intracranial hemorrhage within 36 hours treatment and 2) survive at 90-day post-stroke ,and 3) short hospital length of stay less than 7 days
Improved mRS at discharge | (At discharge) 1 day to 3 months
  Number of patients with improve mRS after treatment at least 1 Score
Improved mRS 3 months | At 3 months
  Number of patients with improve mRS after treatment at least 1 Score
Number of patienta with Length of hospital stay (LOS) less than 7 days Days | 1- 7 days
  Number of patients with LOS < 7 days ( patients must survive )
All complications | 0-4 months
  Number of patients with stroke complications after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assistant Professor Subsai Kongsaengdao, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No